CLINICAL TRIAL: NCT06410222
Title: Risk Factor Analysis and Predictive Models for the Treatment of Recurrent Herpes Zoster Neuralgia Following Short-course Spinal Cord Electrical Stimulation: a Multicenter, Retrospective, Observational Study
Brief Title: Predictive Models for the Treatment of Recurrent Herpes Zoster Neuralgia Following Spinal Cord Electrical Stimulation.
Status: Enrolling by invitation | Type: Observational
Sponsor: Feng Gao (Other)
Collaborators: Shanxi Bethune Hospital (Other); Wuhan No.1 Hospital (Other)
Responsible Party: Sponsor-Investigator, Feng Gao, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-JRB202402013
Record Dates: First submitted 2024-03-27; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Post Herpetic Neuralgia
Keywords: Herpes zoster; post-herpes zoster; spinal cord stimulation
MeSH Terms: conditions — Neuralgia, Postherpetic; Herpes Zoster

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — The diagnostic criteria for pain recurrence at the site of postherpetic neuralgia were numerical rating scale(NRS) score > 4
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Recurrence after undergo spinal cord stimulation — 1. To investigate the pain relief and recurrence of patients with herpes zoster neuralgia after spinal cord stimulation treatment.
  2. To analyze the risk factors related to recurrence after spinal cord stimulation treatment in patients with herpes zoster neuralgia, and build a recurrence prediction model.

SUMMARY:
Shingles is a neuropathic disease caused by varicella-herpes virus(VZV) invading nerves and accompanying pain.Currently, the treatment of postherpetic neuralgia (PHN) includes medication and minimally invasive interventional therapy.In patients with herpes zoster neuralgia treated with spinal cord stimulation (SCS), some patients have satisfactory pain relief after surgery, but some patients have pain symptoms again some time after surgery. The reason for this difference in treatment effect is not clear.

DETAILED DESCRIPTION:
Shingles is a neuropathic disease caused by varicella-herpes virus(VZV) invading nerves and accompanying pain. About 3~5/1000 people suffer from shingles every year in the world, and 2.9~5.8/1000 people over the age of 50 in China suffer from shingles every year, with an annual growth rate of 2.5~5.0%. If acute herpes zoster can not be treated effectively, it will be transformed into postherpetic neuralgia (PHN), patients will suffer long-term knife, needle, burning pain as well as hyperalgesia, touch induced pain and skin paresthesia, which seriously affect the daily life of patients. It also causes a huge social and economic burden.Currently, the treatment of postherpetic neuralgia (PHN) includes medication and minimally invasive interventional therapy. The European Neurological Association has proposed guidelines for first - and second-line drug treatment of herpes zoster neuralgia with level A evidence. At the same time, some patients are relieved by interventional therapy, such as injection therapy (local injection, peripheral nerve block, stellar ganglion block), nerve stimulation therapy (percutaneous electrical nerve stimulation, peripheral nerve stimulation, pulsed radiofrequency), spinal cord stimulation (SCS), and spinal dorsal horn ganglion destruction.

In 1976, spinal cord stimulation (SCS) was first used to treat patients with nociceptive pain. It is to place the stimulation electrode around the diseased nerve for a certain time, frequency, and voltage adjustment, so as to relieve pain. At present, spinal cord stimulation (SCS) has been widely used and studied in the treatment of postherpetic neuralgia (PHN) at home and abroad, and its mechanism of action may be related to the "gate control theory of pain" : in the dorsal horn of the spinal cord, α fiber can inhibit the pain signal transmitted by C fiber, and spinal cord stimulation (SCS) may regulate the transmission of pain signal through this mechanism. At the same time, spinal cord stimulation (SCS) can also affect the levels of gamma-aminobutyric acid and adenosine in the dorsal horn, thereby reducing neuropathic pain.In patients with herpes zoster neuralgia treated with spinal cord stimulation (SCS), some patients have satisfactory pain relief after surgery, but some patients have pain symptoms again some time after surgery. The reason for this difference in treatment effect is not clear. Therefore, this study intends to retrospectively analyze the clinical data of patients with and the risk factors for recurrence after treatment, and then construct a prognostic prediction model to provide evidence and reference for clinical treatment of postherpetic neuralgia (PHN).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old.
* NRS score ≥4 points.
* The pain NRS of previous shingles area treated with SCS was ≤3, and the pain NRS was > 4 after recurrence.

Exclusion Criteria:

* Serious cardiovascular and cerebrovascular diseases, such as heart failure, intracranial aneurysm, hypertension (high risk, very high risk).
* Epilepsy, suffering from mental illness.
* And patients who were lost to follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diagnostic criteria for PHN:
  - In this study, the duration of herpes zoster eruption with pain was greater than or greater than 1 month.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-02-02 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Pain recurrence | up to 1 year
  The diagnostic criteria for pain recurrence at the site of postherpetic neuralgia were Numeric Rating Scales(NRS) score > 4.

SECONDARY OUTCOMES:
The time of electrodes placed in patients | immediately after the surgery
  record the time of spinal cord stimulation in spinal of patients.
Surgical safety indicators | after the surgery 3 days
  record the safety indicators during the spinal cord stimulation surgical ,include the displacement of electrodes and so on.
numeric rating scale(NRS) | After spinal cord stimulation surgical 1 year
  The NRS pain Score is an exponential scale that uses 0 to 10 to represent different levels of pain, 0 being painless and 10 being severe, and asks the patient how bad the pain is, or to circle a number that best represents their pain.
numeric rating scale(NRS) | Day 1 in the hospital
  The NRS pain Score is an exponential scale that uses 0 to 10 to represent different levels of pain, 0 being painless and 10 being severe, and asks the patient how bad the pain is, or to circle a number that best represents their pain.
numeric rating scale(NRS) | the day before the spinal cord stimulation surgical
  The NRS pain Score is an exponential scale that uses 0 to 10 to represent different levels of pain, 0 being painless and 10 being severe, and asks the patient how bad the pain is, or to circle a number that best represents their pain.
C-reactive protein | Day 1 in the hospital
  An according to early infection stricture in serum.When CRP>20mg/l is considered abnormally level .
Albumin | Day 1 in the hospital
  It is a protein that is found in many animal tissues and serum.The normal range 35-50g/L.
diastolic blood pressure | Day 1 in the hospital
  An indicator in blood pressure measurement that indicates the pressure of the heart's arterial blood against the vessel walls during diastole. It is usually measured in millimeters of mercury (mmHg).
systolic blood pressure | Day 1 in the hospital
  A type of blood pressure that refers to the pressure of blood against the artery walls when the heart contracts. It is often used as a measure of cardiovascular health(mmHg).
red blood cell count | Day 1 in the hospital
  The red blood cell count (RBC count) is a measurement of the number of red blood cells present in a microliter (μL) of blood.For males: 4.5 to 5.9 million cells per microliter (μL) of blood.For females: 4.0 to 5.2 million cells per microliter (μL) of blood.
eosinophilic granulocyte | Day 1 in the hospital
  Eosinophils are a type of white blood cell, specifically a subtype of granulocyte, characterized by the presence of eosinophilic granules in their cytoplasm. The normal range for eosinophils is typically between 0% and 6% of the total white blood cell count, though this can vary slightly depending on the laboratory's reference values and the individual's age and health status.
erythrocyte sedimentation rate (ESR) | Day 1 in the hospital
  the sedimentation rate or "sed rate," is a test that measures the rate at which red blood cells (erythrocytes) settle in a tube of blood over a specific period of time.
hemoglobin | Day 1 in the hospital
  Hemoglobin is a protein found in red blood cells that is responsible for transporting oxygen from the lungs to the rest of the body's tissues and organs, and for carrying carbon dioxide back to the lungs for exhalation.The normal range of hemoglobin levels for adult males: 13.8 to 17.2 grams per deciliter (g/dL). adult females: 12.1 to 15.1 g/dL
neutrophilic granulocyte percentage | Day 1 in the hospital
  The neutrophilic granulocyte percentage, often referred to simply as neutrophil percentage or neutrophil count, is a measure of the proportion of neutrophils in the total white blood cell count.a normal neutrophil percentage typically falls within the range of approximately 40% to 75% of the total white blood cell count.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No